CLINICAL TRIAL: NCT06275555
Title: Efficacy and Safety of Bivalirudin Versus Heparin in Anticoagulant Therapy of ECMO: a Randomized Controlled Trial
Brief Title: Use of Bivalirudin for Anticoagulation in Patients With Extracorporeal Membrane Oxygenation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xiaotong Hou (Other)
Responsible Party: Sponsor-Investigator, Xiaotong Hou, Clinical professor, Beijing Anzhen Hospital
Organization: Beijing Anzhen Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2023-101
Record Dates: First submitted 2024-02-17; First posted 2024-02-23 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Extracorporeal Membrane Oxygenation Complication
MeSH Terms: interventions — bivalirudin; Heparin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- bivalirudin group (Experimental): If the creatinine clearance rate > 30ml/min, the initial dose of bivalirudin is 0.04mg/kg/h. If the creatinine clearance rate<30ml/min or the patients who have received renal replacement therapy (CRRT), the initial dose of bivalirudin is 0.02mg/kg/h, and the dose is adjusted according to APPT to maintain APTT at 40-60s. After bivalirudin started, APTT was checked every 4 hours. If APTT was in the target range twice in a row, it was re-examined every 12 hours.
  Interventions: Drug: bivalirudin
- unfractionated heparin group (Other): The initial dose of heparin was 8-12U/kg/h, and the dosage of heparin was adjusted according to the value of APTT. APTT was maintained at 40-60s, and APTT was reexamined every 4 hours.
  Interventions: Drug: unfractionated heparin

INTERVENTIONS:
Drug: bivalirudin — bivalirudin as an anticoagulant
  Arms: bivalirudin group
Drug: unfractionated heparin — unfractionated heparin as an anticoagulant
  Arms: unfractionated heparin group

SUMMARY:
The purpose of this study was to evaluate the efficacy and safety of bivalirudin in anticoagulation therapy in patients with extracorporeal membrane oxygenation (ECMO) compared with unfractionated heparin.

DETAILED DESCRIPTION:
Patients with ECMO who needed systemic anticoagulation were randomly divided into bivalirudin group and unfractionated heparin group;the efficacy of bivalirudin in ECMO anticoagulation was evaluated by comparing the percentage of time within the target anticoagulation level and the incidence of thrombotic complications between the two groups during ECMO; and the safety of bivalirudin in ECMO anticoagulation was evaluated by comparing bleeding complications, blood product infusion and the incidence of acute renal failure between the two groups.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old
2. Accept VA-ECMO or VV-ECMO
3. the ECMO team believes that systemic anticoagulation is necessary and that APTT should be maintained at 40-60s.
4. sign the informed consent form

Exclusion Criteria:

1. previous history of allergy to heparin or bivalirudin
2. previous diagnosis of heparin-induced thrombocytopenia.
3. the pre-random ECMO assistance time is more than 48 hours.
4. pregnant female
5. have participated in this study before.
6. the researchers believe that there are other factors that are not suitable to participate in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Estimated)
Dates: Start 2024-06-03 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
thrombotic complications | Within seven days after starting anticoagulant therapy
  main end point of efficacy
bleeding complications | Within seven days after starting anticoagulant therapy
  main safety endpoint

SECONDARY OUTCOMES:
Hospitalization mortality | 28 days
  All-cause death
Loop replacement | Within seven days after starting anticoagulant therapy
Infusion volume of blood products | Within seven days after starting anticoagulant therapy
  Plasma, platelets and red blood cells
Acute renal failure | Within seven days after starting anticoagulant therapy
  Incidence rate
Heparin-induced thrombocytopenia | Within seven days after starting anticoagulant therapy
  Incidence rate
the time of reaching the target anticoagulant level for the first time | Within seven days after starting anticoagulant therapy
Percentage of time during ECMO within the target anticoagulant level | Within seven days after starting anticoagulant therapy
  APTT maintained at 40-60s

CONTACTS AND LOCATIONS:
Overall Officials: Liangshan Wang, MD, Study Chair — Beijing Anzhen Hospital
Locations (1):
- Beijing Anzhen Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No